CLINICAL TRIAL: NCT04615884
Title: Use of Chinese Herbal Formula Shu Yu Wan in Lung Cancer Patients: a Randomized Double-blind Placebo- Controlled Trial
Brief Title: Use of Chinese Herbal Formula Shu Yu Wan in Lung Cancer Patients
Acronym: CH:II
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to secure the funding despite multiple grant applications
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Thomas Jagoe, Co-Director Peter Brojde Lung Cancer Centre, Jewish General Hospital, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CH:II
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Metastatic NSCLC
Keywords: NSCLC, Metastatic, Symptom management,
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chinese herbs formula: Shu Yu Wan (Experimental): Participants will receive Shu Yu Wan capsules, to take 3 times daily for 6 weeks.
  Interventions: Dietary Supplement: Chinese herbs formula: Shu Yu Wan
- Placebo (Placebo Comparator): Participants will receive capsules to take 3 times daily for 6 weeks.
  Interventions: Other: Placebo capsules

INTERVENTIONS:
Dietary Supplement: Chinese herbs formula: Shu Yu Wan — Shu Yu Wan Formula is a combination of 23 natural chinese herbs.This formula may be used to relieve chemotherapeutic side effects or cancer-related symptoms.
  Arms: Chinese herbs formula: Shu Yu Wan
Other: Placebo capsules — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether Chinese Herb supplements lead to a measurable improvement in symptoms commonly experienced by patients with advanced stage lung cancer and an improvement in quality of life. In our previously conducted single-arm observational study we found significant improvement in physical well-being, tiredness and drowsiness with no evidence of increased toxicity even in those on cytotoxic chemotherapy. Based on the encouraging results of this study we plan to move to a placebo-controlled study using the same Chinese Herb formula.

DETAILED DESCRIPTION:
Despite advances in the design and administration of anti-cancer therapies over recent years, the overall 5-year survival rate for patients with advanced stage lung cancer is 2-4%. These patients frequently suffer a range of different symptoms related to both their disease and it's treatment. As a result, there is a pressing need for research into treatments that may improve their symptoms as well as their quality of life (QOL).

An increasing body of evidence suggests that complementary medicine, including carefully selected combinations of Chinese Herbs (CH), may exert beneficial effects for cancer patients in many ways. The literature suggests that CH combined with chemotherapy can improve survival rates, immediate tumor response, performance status and QOL for those with locally advanced and metastatic disease.

The Shu Yu Wan (SYW) formula used in the feasibility study which demonstrated a significant improvement in symptoms and quality of life will also be employed in this interventional study. THe SYW formula consists of 23 natural Chinese herbs.

This is a randomized, double-blinded, placebo-controlled, parallel-arm clinical trial with a 1:1 allocation ratio for investigating the efficacy and safety of SYW formula for the treatment of lung cancer symptoms. Patients in both groups will receive formula or placebo at a fixed dose for 6 weeks.

After completion of study medication, the treatment will be unblinded and patients randomized to placebo will be offered to cross-over to SYW and will repeat visits Week 0 & Week 6. Patients will be closely monitored for safety and tolerability throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

* Signed informed consent
* Ability to comply with protocol
* Aged ≥18 years
* Histologically or cytologically documented metastatic NSCLC (American Joint Committee on Cancer [AJCC] staging system)
* Prior chemotherapy or radiotherapy is allowed provided the patient has recovered from any toxic effects
* Either off chemotherapy with no plans to start within the next 8 weeks OR on first or second line systemic anti-cancer treatment for NSCLC and completed at least 1 cycle of their current treatment prior to randomization. Permitted chemotherapy regimens are: standard systemic chemotherapy, targeted therapy, immunotherapy or any combinations of the three
* Karnofsky performance status of ≥60
* Life expectancy ≥ 12 weeks
* Adequate hematologic and end-organ function defined by the following laboratory results obtained within 14 days prior to the first study eligibility):

ANC 1. 3 -3.5 x^109/L WBC counts 4.0 - 11 x^109/L Platelet count 150 - 400 x^109/L Hemoglobin 90 -150 g/dL Liver function tests AST ≤ 1.5 x ULN / ALT ≤ 1.5 x ULN L Serum bilirubin 3.0-17.0 x U/L INR ≤1.5 x ULN Creatinine clearance 50-120 mL/min

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study entry:

* Active or untreated central nervous system metastases
* Uncontrolled pleural effusion
* Patients or families who do not speak English or French
* Abnormal liver function as defined above
* Taking regular anti-convulsants, Coumadin or related anti-coagulant
* Taking regular immunosuppressive medications: azathioprine (Imuran), basiliximab (Simulect), cyclosporine (Neoral, Sandimmune), daclizumab (Zenapax), muromonab-CD3 (OKT3, Orthoclone OKT3), mycophenolate (CellCept), tacrolimus (FK506, Prograf), sirolimus (Rapamune), or other immunosuppressive or anti-coagulant that metabolized by liver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Physical Well-Being Scores at Baseline and 6 Weeks | Baseline and 6 weeks
  The primary objective is to compare the change in patient reported Physical Well-Being (PWB) subscale of the Functional Assessment of Cancer Therapy-Lung (FACT-L) questionnaire. The Physical well-being (PWB) subscale has 7 questions with the range of the score from 0 to 4 each. The range of the total score is 0 to 28. The higher the score the better the physical well-being.

SECONDARY OUTCOMES:
Fatigue scores at Baseline and 6 weeks | Baseline and 6 weeks
  The secondary objective is to compare change in Fatigue subscale on the Functional Assessment of Chronic Illness Therapy- Fatigue (FACIT-F) questionnaire. Symptoms and health status will be assessed using the Functional Assessment of Cancer Therapy-lung (FACT-L), and Functional Assessment for Chronic Illness Therapy - Fatigue (FACIT-F). The FACT-L is a 36-item self-report questionnaire that evaluates quality of life in lung cancer patients. Twenty-nine items measure physical, social, emotional and functional well-being; The final 7 items constitute the Lung Cancer Symptom Scale (LCSS). The FACIT-F Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued).

CONTACTS AND LOCATIONS:
Locations (1):
- Peter Brojge Lung Cancer Center, Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Publication in peer-reviewed journal
Supporting Information: Study Protocol, SAP, ICF
Time Frame: March 2024, For 10 years.
Access Criteria: 1. Kasymjanova G, Tran AT, Cohen V, Pepe C, Sakr L, Small D, Agulnik JS, Jagoe RT: The use of a standardized Chinese herbal formula in patients with advanced lung cancer: a feasibility study. Journal of integrative medicine 2018, 16(6):390-395.
URL: https://www.ncbi.nlm.nih.gov/pubmed/30292672